CLINICAL TRIAL: NCT02410564
Title: Testing an Accessible Cognitive Behavioral Therapy for Insomnia (CBT-I) Intervention in Newly Diagnosed Cancer Patients
Brief Title: CBT-I Intervention for Insomnia in Newly Diagnosed Cancer Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: insufficient staff
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Massey Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: MCC-14-10761; HM20002827
Record Dates: First submitted 2015-03-11; First posted 2015-04-07 (Estimated); Last update posted 2016-02-10 (Estimated); Status verified 2016-02

CONDITIONS: Cancer; Chronic Insomnia
Keywords: insomnia; Sleep; CBT-I intervention; SHUTi
MeSH Terms: conditions — Neoplasms; Sleep Initiation and Maintenance Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CBTI treatment (Active Comparator): cognitive behavioral therapy for insomnia (CBTI) treatment is a validated web based version of CBT-I, which will take place over seven weeks and will include a combination of face-to-face and telephone sessions, and email updates
  Interventions: Behavioral: cognitive behavioral therapy for insomnia (CBTI)
- Waitlist control condition (Placebo Comparator): No advice regarding sleep will be given to the control group and if participants ask, they will be informed that such advice can be provided in a few weeks if they choose to crossover to the treatment condition at the end of the study.
  Interventions: Behavioral: Waitlist control condition

INTERVENTIONS:
Behavioral: cognitive behavioral therapy for insomnia (CBTI) — SHUTi program is made up of six, weekly treatment Cores modeled after weekly facetoface(CBTI). Each Core begins by providing a rationale for learning the material, explains main content, homework page with suggestions for improving sleep, and a summarized review of main points. The main content each Core addresses myths about sleep, indepth information about topics, vignettes, and quizzes to evaluate users learning in an interactive. As well as being interactive, SHUTi allows for personalization.Modifications are made to sleep recommendations based in sleep diary data and individually set treatment goals. The cores include Overview, Sleep Behavior Core, Sleep Behavior Core 2, Sleep Education Core, Sleep Thoughts Core, and Problem Prevention Core. Each Core takes approximately 45 to 60 minutes to complete. Cores are presented one at a time; next Core becomes available to users a week after they complete one Core.
  Other Names: SHUTi
  Arms: CBTI treatment
Behavioral: Waitlist control condition — Phone calls with control participants, no advice regarding sleep will be given and if participants ask, they will be informed that such advice can be provided in a few weeks if they choose to crossover to the treatment condition at the end of the study.
  Other Names: control
  Arms: Waitlist control condition

SUMMARY:
To determine the efficacy of a CBT-I intervention in improving sleep and other quality of life outcomes during cancer treatment. To assess the feasibility and acceptability of a CBT-I intervention among newly diagnosed cancer patients.

DETAILED DESCRIPTION:
The proposed study will be a randomized controlled trial design. Participants will be randomized to either a CBTI treatment or a wait list control condition. The intervention is SHUTi, a validated web based version of CBTI, which will take place over seven weeks and will include a combination of face to face and telephone sessions, and email updates. All participants will have a face to face meeting with the doctoral student at enrollment. During the intervention period, all participants will be contacted by telephone at week 1, 3, and 6 to check in and to encourage participant engagement. However, during phone calls with control participants, no advice regarding sleep will be given and if participants ask, they will be informed that such advice can be provided in a few weeks if they choose to crossover to the treatment condition at the end of the study. Participants in SHUTi will additionally be provided the the doctoral student's phone number and will be encouraged to contact her if they have any questions during the intervention. They will also have the option of setting up appointments for face to face meetings during a clinic appointment if they desire additional therapist guidance. Pretreatment, all participants will complete a two week sleep diary and multiple self report measures. At the end of the intervention, all participants will complete a two week sleep diary and multiple self report measures again.

ELIGIBILITY:
Inclusion criteria:

* newly diagnosed with I-III non-metastatic cancer
* scheduled to begin chemotherapy or radiotherapy
* chemotherapy or radiotherapynaïve
* meet diagnostic criteria for chronic insomnia (i.e., lasting for at least one month)
* Chronic insomnia has been defined in previous research:as the presence of (1) three or more episodes of insomnia (i.e., ≥ 30minuteSOL, ≥ 60minute wake after sleep onset (WASO), or ≤ 6.5 hour total sleep time (TST) per night) of per week and (2) daytime effects of insomnia, such as irritability, difficulty concentrating, or fatigue for at least one month.
* interested in behavioral sleep treatment
* have the permission of their oncologists to participate.

Exclusion criteria:

* untreated alcohol or substance abuse or dependence, bipolar, or psychotic disorder
* medical conditions such as seizure disorder, restless leg disorder, or Parkinson's disease
* untreated sleep disorders such as sleep apnea

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2014-12; Primary Completion 2015-07 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
To determine the efficacy of a CBT-I intervention that improves sleep and quality of life outcomes during cancer treatment. | 1 year
  CBT-I is a cognitive behavioral therapy for insomnia. Pretreatment,all participants will complete a two week sleep diary and multiple self report measures. At the end of the intervention, all participants will complete a two week sleep diary and multiple self report measures again.

SECONDARY OUTCOMES:
To assess the feasibility of a CBT--I intervention among newly diagnosed cancer patients. | 1 year
To assess the acceptability of a CBT--I intervention among newly diagnosed cancer patients. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Rybarczyk, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia, United States

REFERENCES:
- [Derived] Cai Z, Tang Y, Liu C, Li H, Zhao G, Zhao Z, Zhang B. Cognitive behavioural therapy for insomnia in people with cancer. Cochrane Database Syst Rev. 2025 Oct 31;10(10):CD015176. doi: 10.1002/14651858.CD015176.pub2. PMID 41170811